CLINICAL TRIAL: NCT02295774
Title: Effect of Oral Administration of Methylene Blue MMX Tablets on Double-stranded DNA Damage Assessed by GammaH2AX Analysis of Colon Biopsy Samples
Brief Title: Effect of Oral Administration of Methylene Blue MMX Tablets on Double Stranded DNA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cosmo Technologies Ltd (Industry)
Responsible Party: Sponsor
Organization: CosmoTech (Unknown)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CB-17-01/08; 2013-000634-35 (EudraCT Number)
Record Dates: First submitted 2014-11-12; First posted 2014-11-20 (Estimated); Results first posted 2016-01-13 (Estimated); Last update posted 2018-11-05 (Actual); Status verified 2018-04

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (Placebo Comparator): Biopsy samples collected during standard white light colonoscopy.
  Interventions: Procedure: standard white light colonoscopy-equivalent to placebo
- Group B (Active Comparator): Subjects who have had samples collected during a Group A colonoscopy, who require a second colonoscopy within 2 weeks. Prior to this second colonoscopy the subjects take Methylene Blue MMX tablets. Biopsies collected are compared to their previous group A colonoscopy for histone gamma H2AX activity.
  Interventions: Drug: Methylene Blue MMX tablets

INTERVENTIONS:
Procedure: standard white light colonoscopy-equivalent to placebo — standard white light colonoscopy
  Arms: Group A
Drug: Methylene Blue MMX tablets — 8x25mg methylene blue MMX tablets administered before a colonoscopy
  Arms: Group B

SUMMARY:
Single Centre, open label assignment phase II clinical study.

To evaluate the effect of oral 200mg Methylene Blue tablets (administered 8x25mg) prior to endoscopy on double stranded DNA breaks in colonic biopsy samples assessed by histone gamma H2AX analysis, compared to control biopsies.

DETAILED DESCRIPTION:
Primary Objective: To evaluate the effect of oral 200 mg Methylene Blue MMX® tablets, (administered as 8 x 25 mg), prior to endoscopy, on double-stranded DNA breaks in colonic biopsy samples assessed by histone γH2AX analysis, compared to control biopsies collected during standard white light colonoscopy without the prior use of Methylene Blue MMX®.

Secondary Objectives : To evaluate the safety and tolerability of oral Methylene Blue MMX® tablets.. To evaluate the staining score for colonoscopy obtained with oral Methylene Blue MMX® tablets . Time to reach the caecum during colonoscopy and withdrawal time from caecum to exit.

ELIGIBILITY:
Inclusion Criteria:

* Males or females, aged between 18 and 75.
* Outpatients scheduled for screening or surveillance colonoscopy
* Subjects must be identified as having the clinical requirement for second colonoscopy within 2weeks of the initial colonoscopy.
* Women of childbearing potential must use at least one reliable method of contraception, be surgically sterilised or be abstinent.
* For female subjects, a negative serum pregnancy test is required before Methylene Blue MMX® tablets are dispensed to the subject.
* Post menopausal patients need to have a period of greater than 1year since last menstrual period.
* Subjects must be able to comprehend the full nature and purpose of the study, including possible risks and side effects.
* Subjects must be able to co-operate with the investigator and to comply with the requirements of the entire study.
* Signed written informed consent prior to inclusion in the study.

Exclusion Criteria:

* No Pregnant or lactating women, or women undergoing fertility treatment.
* No previous medical history of, or suspected hypersensitivity to the Methylene Blue and/or this formulations ingredients.
* No previous medical history of, or suspected hypersensitivity to the PEG based bowel cleansing preparation and/or this formulations ingredients.
* No previous medical history of gastrointestinal obstruction or perforation, toxic megacolon, major colonic resection, severe diverticulitis, heart failure (Class III or IV), serious cardiovascular disease.
* No ALT, AST, GGT, Bilirubin, Creatinine or Urea greater than 2.5 x the upper limit for normal, based on local laboratory testing.
* No clinical alarm symptoms or history of anaemia (previously recorded haemoglobin of less than 10mg/dL) or frank blood in the stool within the last 30 days prior to enrolment.
* No known deficiency of glucose-6-phosphate dehydrogenase.
* No known deficiency of NADPH reductase.
* No treatment within 5 weeks prior to randomisation with Fluoxetine (Prozac).
* No concurrent treatment, or previous treatment within 2 weeks with any of the prohibited psychiatric medications that may interact with Methylene Blue as listed in the Prohibited Medications section; Selective Serotonin Reuptake Inhibitors (SSRI), Serotonin-Norepinepherine Reuptake Inhibitors (SNRI's), listed Tricyclic anti-depressants or Monoamine oxidase A inhibitors.
* No concurrent treatment with anticoagulants, or antiaggregants, inducing an INR > 1.5.
* No current enrolment in any other clinical trial, or previous enrolment in a clinical trial within the last 30 days.
* No other medical condition that in the investigators opinion would make the administration of the study drug or procedures hazardous to the subject.

Exclusion Criteria:

-

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2013-02; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Repici, MD, Principal Investigator — IRCCS Instituto Clinico Humanitas
Locations (1):
- IRCCS Instituto Clinico Humanitas, Rozzano, Italy

REFERENCES:
- [Derived] Repici A, Ciscato C, Wallace M, Sharma P, Anderloni A, Carrara S, Di Leo M, Hassan C. Evaluation of genotoxicity related to oral methylene blue chromoendoscopy. Endoscopy. 2018 Oct;50(10):1027-1032. doi: 10.1055/a-0630-1004. Epub 2018 Jun 15. PMID 29906809

RESULTS

PARTICIPANT FLOW:
Groups:
- MB MMX 200mg: Subjects who have had samples collected during initial colonoscopy, who require a second colonoscopy within 2 weeks. Prior to initial colonoscopy the subjects take 200mg Methylene Blue MMX tablets.
  Biopsies collected are compared to their initial colonoscopy for histone gamma H2AX activity.
  Methylene Blue MMX tablets: 8x25mg methylene blue MMX tablets administered before a colonoscopy
Period: Overall Study
Arm/Group | MB MMX 200mg
Started | 13
Completed | 10
Not Completed | 3
Not completed — Physician Decision | 1
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Population: 13 patients were enrolled. 2 withdrew consent. 1 deviated from inclusion criteria.
  Analysis populations were:
  Analysis set N. subjects
  Safety set 10 FAS 10 PP set 10
  Analysis sets only include those that took the IMP
Groups:
- MB MMX 200mg: Subjects who have had samples collected during initial colonoscopy, who require a second colonoscopy within 2 weeks. Prior to this second colonoscopy the subjects take Methylene Blue MMX tablets. Biopsies collected are compared to their initial colonoscopy for histone gamma H2AX activity.
  Methylene Blue MMX tablets: 8x25mg methylene blue MMX tablets administered before a colonoscopy.
  Subjects were counted as part of an analysis group once they had received the IMP. The discontinued subjects in this study we discontinued before received the IMP.
Arm/Group | MB MMX 200mg
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.1 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 7
Region of Enrollment [Number; unit: participants]
  Italy | 10
Body weight [Mean (Standard Deviation); unit: kg] | 74.40 (15.48)
Height [Mean (Standard Deviation); unit: cm] | 168.2 (11.2)

OUTCOME MEASURES:

1. Primary Outcome: Gamma H2AX Histone Levels in Colonic Biopsy During Standard White Light Colonoscopy and Colonoscopy for Which Methylene Blue MMX Was Taken Prior to Initiating the Colonoscopy
Description: Assay of gamma H2AX histone phosphorylation in biopsy samples collected during colonoscopy.
Time Frame: 2 weeks
Population: FAS = 10
Measure: Number; unit: subject biopsies that tested + for γH2AX
Groups:
- MB MMX 200mg: Subjects who have had samples collected during initial colonoscopy, who require a second colonoscopy within 2 weeks. Prior to this second colonoscopy the subjects take Methylene Blue MMX tablets.
  Biopsies collected are compared to their initial colonoscopy for histone gamma H2AX activity.
  Methylene Blue MMX tablets: 8x25mg methylene blue MMX tablets administered before a colonoscopy
Arm/Group | MB MMX 200mg
Number analyzed (Participants) | 10
subject biopsies that tested + for γH2AX | 0
Statistical Analysis 1: Comparison: MB MMX 200mg; The results of the γH2AX analysis were listed and summarised by frequency tables by visit and colonic region. The results were compared between Visit 2 and Visit 1 for each colonic region and overall using the Mc Nemar's χ2 test. In case of the presence of at least one positive colonic region, that visit was to be considered as 'Positive' for the overall γH2AX analysis; Test type: Superiority or Other; Mc Nemar's χ2 test was not applicable because there is no change between visits; Mc Nemar's χ2 test = 0 — Mc Nemar's χ2 test was not applicable because there is no change between visits

2. Secondary Outcome: To Evaluate the Staining Quality Obtained With Oral Methylene Blue MMX® Tablets.
Description: Staining quality (SC) observed in each colonic region, in the FAS set (N=10); mean (±SD) is reported for SC.
  SC is ranked as follows:
  0 no staining
  1. traces (poor traces in colon mucosa)
  2. detectable (at least the 25% of colon mucosa is stained)
  3. acceptable (at least the 50% of colon mucosa is stained)
  4. good (at least the 75% of colon mucosa is stained)
  5. overstained ( the 100% of the colon mucosa is over stained)
Time Frame: During the colonoscopy
Population: Full Analysis Set (FAS): all included subjects, who received at least one dose of the IMP and had at least one biopsy for the evaluation of the level of γH2AX post-enrolment. This analysis set was used for the primary analysis
Measure: Mean (Standard Deviation); unit: Units on a 6 point scale
Arm/Group | MB MMX 200mg
Number analyzed (Participants) | 10
Units on a 6 point scale
  Ascending colon | 2.9 (1.3)
  Transverse colon | 3.2 (0.8)
  Descending colon | 2.7 (1.2)
  Rectosigmoid | 2.2 (1.6)

ADVERSE EVENTS:
Time Frame: Up to two weeks after IMP administration
Groups:
- MB MMX 200mg: Biopsy samples collected during standard white light colonoscopy.
  No study drug was taken prior to initial Colonoscopy (White light only)
  Subjects who have had samples collected during initial colonoscopy, who require a second colonoscopy within 2 weeks.
  Prior to this second colonoscopy the subjects take Methylene Blue MMX tablets. Biopsies collected are compared to their initial colonoscopy for histone gamma H2AX activity.
  Methylene Blue MMX tablets: 8x25mg methylene blue MMX tablets administered before a colonoscopy
Arm/Group | MB MMX 200mg
All-Cause Mortality (participants affected / at risk) | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13
Other Adverse Events (participants affected / at risk) | 8/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MB MMX 200mg (N=13)
Chromaturia (Renal and urinary disorders) | 8 — Abnormal coloration of the urine.
Faeces discoloured (Gastrointestinal disorders) | 4
Headache (Nervous system disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI must send a manuscript to Sponsor prior to its submission for publication. Sponsor will have 60 days after receipt of the manuscript in which to suggest changes. PI will accept to incorporate the publication comments that do not conflict with the reliability of data, with the rights, the safety and welfare of patients. PI retains the right to publish the result of trial in accordance with current legislation with the consent of the Sponsor subject to the rights of intellectual property.